CLINICAL TRIAL: NCT06547775
Title: A Randomized, Double-blind and Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of KN069 in Chinese Male Participants With Obesity or Overweight
Brief Title: A Study to Evaluate Features of KN069 in Participants With Obesity or Overweight
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Alphamab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KN069-A-101
Record Dates: First submitted 2024-08-02; First posted 2024-08-09 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-09

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1: KN069 Dose 1 (Experimental): Participants will receive a single SC KN069 12mg.
  Interventions: Drug: KN069
- Group 2: KN069 Dose 2 (Experimental): Participants will receive a single SC KN069 30mg.
  Interventions: Drug: KN069
- Group 3: KN069 Dose 3 (Experimental): Participants will receive a single SC KN069 60mg.
  Interventions: Drug: KN069
- Group 4: KN069 Dose 4 (Experimental): Participants will receive a single SC KN069 120mg.
  Interventions: Drug: KN069
- Group 5: KN069 Dose 5 (Experimental): Participants will receive a single SC KN069 240mg.
  Interventions: Drug: KN069

INTERVENTIONS:
Drug: KN069 — Solution for SC injection

SUMMARY:
This is a Phase 1, First-in-human, double-blinded, placebo-controlled study which aims to investigate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and the immunogenicity of KN069 in Chinese male participants with Obesity or Overweight.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 18-55 years old (including threshold);
2. Body mass index (BMI)：24.0 kg/m2≤BMI<35 kg/m2；
3. HbA1c<6.5%；3.9mmol/L≤Fasting blood glucose level <7.0mmol/L；
4. Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures and are willing to follow study restrictions; Are able and willing to sign the ICF.

Exclusion Criteria:

1. Those who have a history of chronic diseases or are currently suffering from obvious systemic diseases, such as diseases of cardiovascular system, respiratory system, endocrine and metabolic system, urinary system, digestive system, blood system, autoimmune system, neurological or psychiatric system, bacterial or viral infection;
2. History of acute or chronic pancreatitis; A personal or family history of medullary thyroid cancer or multiple endocrine adenoma syndrome type 2; A history of other malignancies;
3. History of GI disorder (for example, relevant esophageal reflux or gall bladder disease) or any GI disease which impacts gastric emptying (for example, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by GLP-1 analogs or DPP-IV inhibitors;
4. Participants had cholecystolithiasis (removal of gallstones) or cholecystectomy (removal of gall bladder) in the past;
5. Allergies to KN069 excipients or drugs similar to KN069 in structure or KN069 in the same category;
6. A history of medicine abuse/dependence or narcotics abuse within 1 year prior to the screening and/or show positive findings on urinary drug screening;
7. Have undergone any major surgery or surgery affecting drug absorption, distribution, metabolism, excretion within the 3 months prior to screening, or are scheduled to undergo surgery during the trial period (major surgery is defined as surgery on the intracranial, chest, abdomen, pelvic, or limb organs that result in major tissue trauma and require long-term recovery).
8. Drinking more than 14 units of alcohol per week (1 unit =360ml beer or 45ml liquor with 40% alcohol or 150ml wine) in the 3 months before or during the screening period, alcohol cannot be banned during the hospital stay, and alcohol consumption cannot be limited to less than 2 units of alcohol per day during the post-discharge visit.
9. Blood donation or blood loss ≥ 300 mL within 3 months prior to screening, or blood/blood components donation planned during the trial or within 1 month after the final study visit.
10. Received administration of other drugs/vaccines in clinical trials within 2 months prior to screening; In other clinical trials at the time of screening;
11. People who diet or undergo weight loss treatment within 2 months (for whatever reason) before administration, or who have made significant changes in their lifestyle habits.;
12. Received vaccination within 14 days prior to screening, or have vaccination schedule during the trial, including inactivated vaccine, live attenuated vaccine, recombinant protein vaccine, recombinant adenovirus vaccine, RNA vaccine, DNA vaccine, COVID-19 vaccine;
13. Use medication (including prescription drugs, over-the-counter drugs, herbal medicine) with the exception of vitamin/mineral supplements, paracetamol, topical medication, and contraceptives within 14 days prior to dosing.
14. Use of GLP-1 analogues, GLP-1 receptor agonists, or any other formulations related to incretin and other drugs that the investigator believes may affect the trial within the 3 months prior to administration.
15. Any abnormal patients who met the following criteria during screening: 1) serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) exceeded the upper limit of the reference value range by 2 times; Serum total bilirubin (TBIl) exceeded 1.5 times the upper limit of the reference value range; 2) Fasting triglyceride (TG) ≥5.6mmol/L; 3) Physical examination, vital signs, electrocardiogram, laboratory examination, imaging and other abnormalities have clinical significance, and the investigator judges that they may pose a major risk to the subjects or interfere with the evaluation of safety, PK or PD results and are not suitable to participate in the trial;
16. Positive breath test for alcohol (>0 mg/100 mL);
17. Evidence of hepatitis B/hepatitis C/HIV/syphilis.
18. Urine screen positive for drug abuse.
19. Participants that refuse to stay abstinent, and refuse to consistently use a form of highly effective birth control method starting at Screening (signing the ICF) and continuing throughout the clinical study period, and to 3 months after administration of IP; or to have a birth plan during the screening period until 3 months after dosing;
20. Participants that plan to donate sperms from dosing until 3 months after administration of IP.
21. Due to trauma, surgery, allergies or skin lesions, the abdominal skin is not suitable for subcutaneous injection.
22. Other factors that the investigator considers unacceptable for participation in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | Up to Day 42

SECONDARY OUTCOMES:
To evaluate the plasma concentration of KN069 | Up to Day 42
To evaluate the Area under the plasma concentration versus time curve (AUC) of KN069 | Up to Day 42
To evaluate the weight (kg) change from baseline | Up to Day 42
To evaluate the waist circumference (cm) change from baseline | Up to Day 42
To evaluate the BMI (kg/m^2) change from baseline | Up to Day 42
Number of Participants with Anti-KN069 Antibodies | Up to Day 42

CONTACTS AND LOCATIONS:
Overall Officials: GuoPing Yang, Doctor, Principal Investigator — Xiangya Third Hospital, Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided